CLINICAL TRIAL: NCT05810142
Title: Clinical Study on Third-line Treatment of Advanced Duodenal Adenocarcinoma by Fuquinitinib Combined With Sindillimab
Status: Not yet recruiting | Type: Observational
Sponsor: RenJi Hospital (Other)
Responsible Party: Principal Investigator, chengxiaojiao, Attending physician, RenJi Hospital
Other Study IDs: RJ-FC-ADA-1
Record Dates: First submitted 2023-03-30; First posted 2023-04-12 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-03

CONDITIONS: Third-line Treatment; Dvanced Duodenal Adenocarcinoma; Furquinelone Combined With Sintilimab
MeSH Terms: interventions — sintilimab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: furquimatinib and sintilimab — furquimatinib and sintilimab

SUMMARY:
This research project is a single-center, retrospective clinical exploration study. It aims to retrospectively analyze data from 20 patients with advanced duodenal adenocarcinoma who received third-line treatment with furquinelone combined with sintilimab, in order to determine the clinical efficacy and safety of this combination therapy in advanced duodenal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients must meet all of the following criteria to be eligible for inclusion:

Age between 18 and 80 years (inclusive); Imaging findings consistent with unresectable local advanced, recurrent or metastatic duodenal adenocarcinoma; Histologically confirmed unresectable local advanced, recurrent or metastatic duodenal adenocarcinoma; ECOG performance status 0-2; At least one measurable or evaluable lesion according to RECIST v1.1; Third-line or above treatment with the combination of sintilimab and furquimatinib.

Exclusion Criteria:

-

Patients meeting any of the following criteria will be excluded:

Patients with incomplete clinical data or laboratory examination that affects statistical analysis; Patients who have had other malignant tumors in the past 5 years; Patients who have had arterial thrombotic diseases such as angina, myocardial infarction, and transient ischemic attack in the past 6 months; Patients who have received other types of anti-tumor or experimental treatment; Pregnant or lactating women; Patients with other diseases or abnormal mental status that may affect the patient's treatment; Patients who have received other types of immune therapy, anti-angiogenic drugs, or small-molecule tyrosine kinase inhibitors.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will include patients with advanced duodenal adenocarcinoma who received third-line or above treatment with the combination of furquimatinib and sintilimab in Renji Hospital from January 2019 to the present.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Primary efficacy endpoint: Objective Response Rate (ORR) | 2 years

IPD SHARING:
Plan to Share IPD: Undecided